CLINICAL TRIAL: NCT03689127
Title: Influence of Heated Breathing Circuit on Postoperative Sore Throat in Patients Undergoing Double-lumen Endobronchial Tube Insertion
Brief Title: Heated Breathing Circuit on Postoperative Sore Throat After Double-lumen Endobronchial Tube Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Heated Circuit POST
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Lung Surgery
Keywords: intubation; pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Heated breathing circuit will be turned off.
  Interventions: Device: Heated breathing circuit off
- Heat (Experimental): Heated breathing circuit will be turned on.
  Interventions: Device: Heated breathing circuit on

INTERVENTIONS:
Device: Heated breathing circuit on — Heated breathing circuit will be turned on.
  Arms: Heat
Device: Heated breathing circuit off — Heated breathing circuit will be turned off.
  Arms: Control

SUMMARY:
This investigation is planned to compare the incidence and severity of postoperative sore throat according to the use of heated breathing circuit in patients undergoing double-lumen endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for double-lumen endotracheal intubation

Exclusion Criteria:

* Difficult airway
* Mallampatti scores greater than 2
* Recent sore throat
* Cervical spine disease
* Recent upper respiratory infection
* Recent analgesics
* History of head and neck surgery
* Friable teeth
* Multiple intubation attempts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative sore throat for postoperative 24 h | At 24 hours

SECONDARY OUTCOMES:
Number of participants with postoperative sore throat | At 1, 6, and 24 hours
Postoperative sore throat scores | At 1, 6, and 24 hours
Number of participants with postoperative hoarseness | At 1, 6, and 24 hours
Number of participants with postoperative shivering | At 1, 6, and 24 hours
Wound pain scores | At 1, 6, and 24 hours
  Visual anlogue scales will be used (10: most imaginable pain, 0: no pain).
Jaw discomfort scores | At 1, 6, and 24 hours
  Visual anlogue scales will be used (10: most imaginable pain, 0: no pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Hyun-Chang Kim, Daegu, Non-US/Canada, South Korea

IPD SHARING:
Plan to Share IPD: Undecided